CLINICAL TRIAL: NCT05516745
Title: E-monitoring of Pulmonary Function in Patients With Duchenne Muscular Dystrophy Undergoing Respiratory Rehabilitation at Home"
Brief Title: E-monitoring of PULMonary Function in Patients With Duchenne Muscular Dystrophy at Home"
Acronym: E-PULMoDMD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: EPULMoDMD 001/2021
Record Dates: First submitted 2021-09-22; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
Keywords: AioCare spirometer; home spirometry; spirometry e-monitoring; pulmonary rehabilitation; digital medicine; e-health
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Intervention Model Description: 4 arms -
  1. arm - AioCare device spirometry
  2. arm - AioCare device spirometry+ telerehabilitation of the respiratory system
  3. arm - telerehabilitation of the respiratory system
  4. arm - control arm - standard of care (no monitoring, no telerehabilitation)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- arm with intervention (AioCare spirometry) (Experimental): 50 participants with DMD aged 7-17 years, subjected to home electronic monitoring
  Interventions: Device: AioCare spirometer
- arm with intervention (AioCare spirometry with telerehabilitation) (Experimental): 50 participants with DMD aged 7-17 years, subjected to home electronic monitoring with the AioCare device and pulmonary rehabilitation exercises
  Interventions: Device: AioCare spirometer; Other: telerehabiliation of the respiratory system
- arm with intervention (telerehabilitation) (Experimental): 50 participants with DMD aged 7-17 years, subjected to pulmonary rehabilitation exercises
  Interventions: Other: telerehabiliation of the respiratory system
- control arm (no intervention) (No Intervention): 50 participants with DMD aged 7-17 years, subject to a standard of care

INTERVENTIONS:
Device: AioCare spirometer — In the first part of the trial, all participants from arms 1 and 2 will receive the AioCare spirometer (Healtup, Poland) to home-based monitoring pulmonary function. Hospital spirometry examinations (Jaeger, Germany) evaluating disease progression will be performed periodically. There are to be follow-up visits after 3 months and after 6 months. The end-point visit is planned for 12 months.
  Arms: arm with intervention (AioCare spirometry with telerehabilitation); arm with intervention (AioCare spirometry)
Other: telerehabiliation of the respiratory system — A major component of respiratory dysfunction seems to be a decline of respiratory muscle weakness. The proposition is respiratory telerehabilitation to improve the function of respiratory muscles. Telerehabilitation includes breathing exercises for use at home. The participants will be trained in the hospital and will receive video presentations to support the exercises at home.
  Arms: arm with intervention (AioCare spirometry with telerehabilitation); arm with intervention (telerehabilitation)

SUMMARY:
Duchenne muscular dystrophy (DMD) is the most common, progressive, irreversible muscular dystrophy. The pulmonary function is crucial for the duration of life in this disease. The European Respiratory Society is currently focused on digital health, seeking to define the realistic innovations for digital respiratory medicine to support professionals and patients during the COVID-19 pandemic. This study aimed to investigate whether it is possible to monitor pulmonary function at home by using an individual electronical spirometry system in children with Duchenne muscular dystrophy DMD. The second aim of the study is the implementation of respiratory telerehabilitation and the assessment of its impact on pulmonary function (FVC).

DETAILED DESCRIPTION:
Duchenne muscular dystrophy (DMD) is the most common muscular dystrophy. DMD is a genetically determined, progressive, irreversible disease in which dystrophin dysfunction in skeletal and multiple organ muscles is fatal before the age of 20 years. Respiratory muscle failure is the most common cause of death.

In the first years of life, the respiratory system of children with DMD is efficient and does not differ from that of healthy peers. From the age of 7 years, the parameters of lung function no longer increase, and between the ages of 10 to 12 years, when the child loses the ability to walk independently, the lung function rapidly deteriorates.

Currently, it is not possible to cure the disease, but appropriate medical management may improve the quality of life and prolong the survival of patients with DMD.

The basic tasks include the initiation of early monitoring of respiratory system functions. It is recommended that measurement of lung function is started from the age of 5 years. Taking the measurement at such an early age is aimed at familiarizing and teaching the child about this type of systematic examination and determining the individual maximum parameters of lung function in each child. Thanks to systematic measurements, it is possible to detect any sharp deterioration as well as the moment when the decreasing lung function requires respiratory support, so-called non-invasive ventilation (NIV).

According to the standards, lung function is assessed by spirometry, which should be performed at least once a year, at least every 6 months after losing independent walking, and every 3 months after starting non-invasive ventilation.

The spirometry test assesses forced vital capacity (FVC), which is considered a marker of disease progression. An FVC value below 2.1 L is a rationale to start supporting the cough reflex, and below 1 L is an indication to start respiratory support, i.e. NIV.

Implementation of the above-mentioned tests often encounters difficulties that increase when the child loses independent walking. Additionally, during the COVID pandemic, spirometry was included in the procedures generating aerosols, i.e. high risk of SARS-CoV-2 virus transmission. Therefore, it has become necessary to look for other methods of measuring and monitoring lung function in children with DMD.

The presented project aims to evaluate the measurement of lung function at home using an individual spirometer called an AIOCARE.

The AioCare spirometer is a small, convenient device that can be used anywhere. The device enables systematic non-invasive monitoring of lung parameters (including FVC measurement) at home in children over 5 years of age. The child inhales and exhales forcefully through a mouthpiece with antibacterial and antiviral filters. The test results are sent from the AioCare spirometer via the AioCare application for iOS and Android (as used by all current smartphones). Communication between the AioCare spirometer and the application takes place via a Bluetooth 4.0 (BT LE) connection. The spirometry results are available to the practitioner in real-time in the AIOCARE Doctor panel.

Additionally, a module with exercises for training respiratory muscles, included in an additional smartphone application, will be added to the daily spirometry test as part of the project.

It will be a series of 4 exercises aimed at strengthening respiratory muscles, to be performed before the spirometry test.

The assumption of the exercises is the possibility of performing them independently, at home, without the assistance of a physiotherapist, and without the use of additional equipment. Participants will perform forced exhalation exercises with a relaxed epiglottis, exercises to improve the mechanics of the chest and the mobility of the shoulder girdle. The exercises will be performed each day. The duration of the exercises is approximately 7 minutes. The exercise program will be recorded in the form of an instructional video.

Pulmonary rehabilitation is one of the key issues in DMD patient management. The combination of systematic lung function measurement with home respiratory rehabilitation is an innovative project. It is a non-invasive test, and the measurement is intended to improve the quality of life of DMD patients.

Aims of the study:

1. to assess pulmonary function for 12 months using home electronic monitoring (AioCare System) in DMD participants aged 7-18 years (number of participants with increase FVC %pv, L value).
2. to assess the acceptance of electronic home monitoring of a respiratory system in this group of patients (number of participants accepted home e-monitoring, survey).
3. to compare the results from home electronic spirometry (AioCare) with results from hospital spirometry (Jaeger, Germany) - (value of FVC%pv, L).
4. to investigate whether it is possible to conduct respiratory physical therapy with the use of telerehabilitation in DMD patients (number of patients accepted telerehabilitation, survey).
5. to evaluate the impact of home telerehabilitation on pulmonary function (number of patients with increased FVC%pv, L value)
6. to assess the quality of life of patients subjected to electronic monitoring and pulmonary rehabilitation vs. not subjected

Study group: 200 participants with DMD aged 7-18 years, in the 4 arms (50 participants each): (1) subjected to home electronic monitoring exercises with the AIOCARE device, (2) home electronic monitoring with AioCareand pulmonary rehabilitation; (3) telerehabilitation of respiratory system; (4) control group - no interventions.

Duration of the project March 2021 - March 2025.

ELIGIBILITY:
Inclusion Criteria:

* male, ≥7 years and <18 years of age at the time of enrollment in the study;
* ability to perform spirometry;
* stated willingness to comply with all study procedures and availability for the duration of the study.

Exclusion Criteria:

* no consent to participate in the study;
* patients under 7 years of age or above 18 years of age;
* inability to perform spirometry

Ages: 7 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2021-03-20 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline of the mean Forced Vital Capacity in Liters measured by home and hospital spirometry in DMD participants with vs without respiratory telerehabilitation | 12 months
  Some studies showed that respiratory function declines at a rate of 6-11% annually in patients with DMD. A major component of respiratory dysfunction seems to be a decline of inspiratory muscle weakness. Methods of improving the functioning of the muscles of the respiratory system are constantly sought. One of the key factors that can improve the function of respiratory muscles is proper rehabilitation. The proposition is implementation of telerehabilitation of respiratory muscle together with e-monitoring pulmonary function at home.
Change from Baseline of the mean Forced Vital Capacity in %predicted value measured by home and hospital spirometry in DMD participants with vs without respiratory telerehabilitation | 12 months
  Some studies showed that respiratory function declines at a rate of 6-11% annually in patients with DMD. A major component of respiratory dysfunction seems to be a decline of inspiratory muscle weakness. Methods of improving the functioning of the muscles of the respiratory system are constantly sought. One of the key factors that can improve the function of respiratory muscles is proper rehabilitation. The proposition is implementation of telerehabilitation of respiratory muscle together with e-monitoring pulmonary function at home.

SECONDARY OUTCOMES:
Possibility of home e-monitoring of pulmonary function in patients with Duchenne Muscular Dystrophy in the Covid-19 pandemic | 4 weeks
  * number of the days with performed spirometry test per patient during the monitoring period
  * number and percent of correct spirometry parameters.
The number of the participants who performed at least one correct spirometry examination | 4 weeks
  Feasibility of home e-monitoring of pulmonary function in patients with Duchenne Muscular Dystrophy in the Covid-19 pandemic measured by The number of the participants who performed at least one correct spirometry examination
the difference in the value of spirometry results (FVC %pv, L) between home spirometry and spirometry in the hospital | 4 weeks
  Feasibility of home e-monitoring of pulmonary function in patients with Duchenne Muscular Dystrophy in the Covid-19 pandemic measured by The number of the participants who performed at least one correc the difference in the value of spirometry results (FVC %pv, L) between home spirometry and spirometry in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Eliza Wasilewska, MD,PhD, Principal Investigator — Medical University Gdansk
Locations (1):
- Medical University, Gdansk, Poland

REFERENCES:
- [Result] Birnkrant DJ, Bushby K, Bann CM, Apkon SD, Blackwell A, Brumbaugh D, Case LE, Clemens PR, Hadjiyannakis S, Pandya S, Street N, Tomezsko J, Wagner KR, Ward LM, Weber DR; DMD Care Considerations Working Group. Diagnosis and management of Duchenne muscular dystrophy, part 1: diagnosis, and neuromuscular, rehabilitation, endocrine, and gastrointestinal and nutritional management. Lancet Neurol. 2018 Mar;17(3):251-267. doi: 10.1016/S1474-4422(18)30024-3. Epub 2018 Feb 3. PMID 29395989
- [Result] Birnkrant DJ, Bushby K, Bann CM, Alman BA, Apkon SD, Blackwell A, Case LE, Cripe L, Hadjiyannakis S, Olson AK, Sheehan DW, Bolen J, Weber DR, Ward LM; DMD Care Considerations Working Group. Diagnosis and management of Duchenne muscular dystrophy, part 2: respiratory, cardiac, bone health, and orthopaedic management. Lancet Neurol. 2018 Apr;17(4):347-361. doi: 10.1016/S1474-4422(18)30025-5. Epub 2018 Feb 3. PMID 29395990
- [Result] Finder JD, Birnkrant D, Carl J, Farber HJ, Gozal D, Iannaccone ST, Kovesi T, Kravitz RM, Panitch H, Schramm C, Schroth M, Sharma G, Sievers L, Silvestri JM, Sterni L; American Thoracic Society. Respiratory care of the patient with Duchenne muscular dystrophy: ATS consensus statement. Am J Respir Crit Care Med. 2004 Aug 15;170(4):456-65. doi: 10.1164/rccm.200307-885ST. No abstract available. PMID 15302625
- [Result] Phillips MF, Quinlivan RC, Edwards RH, Calverley PM. Changes in spirometry over time as a prognostic marker in patients with Duchenne muscular dystrophy. Am J Respir Crit Care Med. 2001 Dec 15;164(12):2191-4. doi: 10.1164/ajrccm.164.12.2103052. PMID 11751186
- [Result] Toussaint M, Chatwin M, Soudon P. Mechanical ventilation in Duchenne patients with chronic respiratory insufficiency: clinical implications of 20 years published experience. Chron Respir Dis. 2007;4(3):167-77. doi: 10.1177/1479972307080697. PMID 17711917
- [Result] LoMauro A, D'Angelo MG, Aliverti A. Sleep Disordered Breathing in Duchenne Muscular Dystrophy. Curr Neurol Neurosci Rep. 2017 May;17(5):44. doi: 10.1007/s11910-017-0750-1. PMID 28397169
- [Result] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- See also: AioCare description — https://healthcloud.aiocare.com

DOCUMENTS (1):
  • Study Protocol (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT05516745/Prot_000.pdf